CLINICAL TRIAL: NCT02733198
Title: Effect of a Prognostic Algorithm to Reduce Length of Stay in Acute Pulmonary Embolism: a Randomized Controlled Trial
Brief Title: Prognostication in Acute Pulmonary Embolism
Acronym: IPEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Spain (Other Government)
Responsible Party: Principal Investigator, David Jimenez, Pulmonary physician, Ministry of Health, Spain
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PI15/00207
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prognosis-guided (Experimental): Duration of bed rest and duration of length of stay will be guided according to a predefined prognostic algorithm.
  Interventions: Other: Prognosis-guided therapy
- Standard medical therapy (No Intervention): Duration of bed rest and duration of length of stay will be decided by the attending physician.

INTERVENTIONS:
Other: Prognosis-guided therapy
  Arms: Prognosis-guided

SUMMARY:
To evaluate the effect of a prognosis-guided vs standard medical therapy in the: 1) duration of hospital stay; 2) cost-effectiveness; 3) satisfaction and quality of life; 4) in-hospital and 30-day all-cause mortality; and 5) 30-day readmissions in normotensive patients with acute symptomatic pulmonary embolism (PE).

Design: Prospective, randomized, controlled, single blind trial. Normotensive patients with acute symptomatic PE will be randomly assigned to follow a prognosis-guided treatment, or to receive usual care.

Setting: Respiratory, Medicine and Emergency Departments in 15 Spanish hospitals.

Analyses: Data for the primary and secondary end points will be analyzed according to the intention-to -treat principle. The intention-to-treat analysis will include all randomly assigned patients. For the efficacy end points, investigators will use the Mann-Whitney U test. We will also use competing risk regression models according to Fine and Gray. For the safety end points, comparisons will be made with the use of the chi-square test. Separate analyses will be done in key prespecified subgroups of patients, according to age and hospital size.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PE by objective testing
* Signed and dated informed consent of the subject available before the start of any specific trial procedures

Exclusion Criteria:

* Pregnancy
* Haemodynamic instability
* Contraindication to anticoagulant therapy
* Life expectancy less than 3 months
* Participation in other clinical trials during the present clinical trial
* Use of a fibrinolytic agent, surgical thrombectomy, interventional (transcatheter) thrombus aspiration or lysis, or use of a cava filter to treat the index episode of PE
* Inability to the follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 30-days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramon y Cajal, IRYCIS, Alcala de Henares University, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jimenez D, Rodriguez C, Pintado B, Perez A, Jara-Palomares L, Lopez-Reyes R, Ruiz-Artacho P, Garcia-Ortega A, Bikdeli B, Lobo JL; IPEP investigators. Effect of Prognostic Guided Management of Patients With Acute Pulmonary Embolism According to the European Society of Cardiology Risk Stratification Model. Front Cardiovasc Med. 2022 Apr 12;9:872115. doi: 10.3389/fcvm.2022.872115. eCollection 2022. PMID 35497990
- [Derived] Jimenez D, Rodriguez C, Leon F, Jara-Palomares L, Lopez-Reyes R, Ruiz-Artacho P, Elias T, Otero R, Garcia-Ortega A, Rivas-Guerrero A, Abelaira J, Jimenez S, Muriel A, Morillo R, Barrios D, Le Mao R, Yusen RD, Bikdeli B, Monreal M, Lobo JL; IPEP investigators. Randomised controlled trial of a prognostic assessment and management pathway to reduce the length of hospital stay in normotensive patients with acute pulmonary embolism. Eur Respir J. 2022 Feb 10;59(2):2100412. doi: 10.1183/13993003.00412-2021. Print 2022 Feb. PMID 34385269